CLINICAL TRIAL: NCT04771091
Title: Correlation Between Head Perineum Distance Measured by Trans-périneal Ultrasound and Delivery Mode in Patient in the Second Stage of Labor
Brief Title: Head-perineum Distance and Delivery Mode
Acronym: EchoPé
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 35RC20_3011_EchoPé
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Pregnancies; Obstetric Labor
Keywords: Head perineum distance; ultrasound measure; delivery mode; instrumental delivery; spontaneous delivery; pushing maternal efforts
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mesure of head-perineum distance by transperineal ultrasound (Experimental): A mesure of head-perineum distance by ultrasound will be realized at the beginning of maternal pushing efforts by a junior gynecologist.
  Interventions: Diagnostic Test: Mesure of head-perineum distance by transperineal ultrasound

INTERVENTIONS:
Diagnostic Test: Mesure of head-perineum distance by transperineal ultrasound — A mesure of head-perineum distance by ultrasound will be realized at the beginning of maternal pushing efforts by a junior gynecologist
  Other Names: Echography

SUMMARY:
In a prospective cohort of patients in the second phase of labor, the investigators measured the head-perineum distance and correlate it to the mode of delivery (spontaneous delivery - instrumental delivery - ceasarean section).

DETAILED DESCRIPTION:
Head-perineum distance measured by transperineal ultrasound is a simple and well-known tool to help diagnose the fetal head engagement and predictive value to instrumental extraction succeeds.

It is performed in labor room and is a non-invasive test, realized on a healthy skin.

The investigators performed a systematical measure of head perineum distance at the beginning of the expulsive labor phase. The investigators made the hypothesis, based on our clinical experience, that starting expulsive labor phase with head perineum distance greater than forty five millimeters, lead to an increased risk of instrumental extraction and therefore an increase in materno-fetal morbidity and mortality.

The investigators sought to evaluate the optimal head perineum distance at the beginning of expulsive efforts.

ELIGIBILITY:
Inclusion Criteria:

* Single pregnancy
* In labor (spontaneous or induced)
* Term superior at 37 SA
* Delivery by summit presentation

Exclusion Criteria:

* Non single pregnancy
* Suspected malformative abnormalities in the unborn fetus
* Refusal of participation
* Minor patient
* Adult patient subject to legal protection or patient deprived of liberty
* Poor French language understanding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2021-04-04 (Actual); Study Completion 2021-04-04 (Actual)

PRIMARY OUTCOMES:
Delivery mode | Day 1
  spontaneous or instrumental vaginal delivery

CONTACTS AND LOCATIONS:
Overall Officials: Maela Le Lous, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- Centre Hospitalier Universitaire de Rennes, Rennes, France